CLINICAL TRIAL: NCT06961552
Title: The Effect of Reflexology on Premenstrual Syndrome Symptoms, Pain and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Bingöl, MSc, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-DB
Record Dates: First submitted 2025-04-21; First posted 2025-05-08 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Effect of Reflexology on Premenstrual Syndrome Symptoms
Keywords: reflexology; Premenstrual Syndrome-PMS; Pain; Quality of Life
MeSH Terms: conditions — Premenstrual Syndrome; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology massage group (Experimental)
  Interventions: Other: reflexology masaj group
- control group (No Intervention)

INTERVENTIONS:
Other: reflexology masaj group — The women in the reflexology group will receive a reflexology massage with proven regional applications, pressure sliding and circular pressure three times with baby oil for two cycles by the researcher, starting at the end of menstruation (5-7th days of the cycle), for a total of 30 minutes in a single session for each foot, starting at 15 minutes per foot. A total of 8 reflexology massage sessions will be performed, one session per week (Monday) for 8 weeks.
  Arms: reflexology massage group

SUMMARY:
This study was planned as a randomized controlled experimental study to examine the effect of reflexology on premenstrual syndrome symptoms, pain and quality of life in women with premenstrual syndrome between January 2025 and December 2025.

A total of 70 women, 35 in the experimental group and 35 in the control group, who applied to the gynecology outpatient clinic with premenstrual syndrome symptoms, met the inclusion criteria and agreed to participate in the study voluntarily will constitute the sample.

The women in the reflexology group will receive a reflexology massage for two cycles by the researcher, starting at the end of menstruation (on the 5th-7th days of the cycle), for a total of 30 minutes, with proven applications specific to the region, pressure sliding and circular pressure applied to the reflexology distribution points on the foot bones three times, with baby oil. A total of 8 reflexology massage sessions will be performed, one day a week (Monday) for 8 weeks, one session. No intervention will be made to the control group.

DETAILED DESCRIPTION:
The menstrual cycle is defined as a periodic preparation period for fertilization and pregnancy that begins after puberty and continues until menopause. Women may experience some symptoms commonly in the premenstrual and menstrual periods during the menstrual cycle, which is a physiological process.

Premenstrual syndrome is a condition that is seen in the late luteal phase of the menstrual cycle, recurs in most cycles, rapidly improves with menstruation, and is not seen for at least one week in the follicular phase, and in which cognitive, physical, somatic and emotional behavioral changes are observed. PMS symptoms typically begin after the 13th day of the menstrual cycle. It is suggested that it is difficult to determine the true prevalence due to the variety of PMS symptoms. International studies report that the prevalence of PMS varies between 7.1% and 99.5%. Similarly, studies conducted in Turkey report that the prevalence of PMS is between 33-92.3%.

The severity and occurrence of PMS symptoms vary from woman to woman. Physical symptoms seen in PMS are appetite changes, weight gain, nausea, abdominal distension, diarrhea, constipation, breast tenderness, fullness, hot flushes, acne, muscle and joint pain, and headache. Behavioral symptoms are changes in sexual desire, changes in work habits, social withdrawal, avoidance of human relations, crying spells, tendency to fight, apathy, difficulty concentrating, and sleep disorders. Psychological symptoms are forgetfulness, decreased self-esteem, feelings of inadequacy, guilt, paranoia, irritability, anxiety, restlessness, hypersensitivity to sound and light, loneliness, suicidal thoughts, psychosis, confusion, variable and depressive mood, decreased concentration, and a feeling of losing control. PMS also has a very negative effect on women's quality of life. Premenstrual symptoms can lead to increased accident potential and economic losses. It can also negatively affect young girls' emotional well-being, self-confidence, academic success, attendance at classes, work quality, daily activities, social activities, social relations, family relations and quality of life.

Reflexology is a holistic and complementary treatment method. Unlike regular massage, a special pressure technique is used to apply rubbing, patting and squeezing movements to reflex points. The thumb and index finger are mostly used to apply pressure. The International Reflexology Institute defines reflexology as "a technique that is applied manually to reflex points on the hands, feet and ears, which are associated with all glands, organs and body parts, and helps normalize body functions." Reflexology has been used since ancient times to balance the energy in the body, provide healing and increase relaxation.

In recent years, it has been reported that reflexology reduces fatigue, insomnia, stress, anxiety, depression, dyspnea, migraine pain, rheumatic muscle pain and spasm, supports general rehabilitation practices in neurological diseases such as multiple sclerosis, reduces nausea, vomiting and constipation, alleviates some urinary system problems, cancer pain and side effects of chemotherapy, facilitates birth, reduces pain during birth, after birth and after surgery, premenstural syndrome (PMS) and dysmenorrhea complaints, vasomotor problems in menopause, infantile colic and pain in babies, regulates the sedation level and vital signs of patients. The top five issues are pain (28.1%), fatigue (21.9%), anxiety (18.8%), quality of life (15.6%) and sleep quality (12.5%).

Nurses are health professionals who support women with PMS from the first stage of symptom management. Health education is very important in coping with PMS. Education should raise awareness that menstruation is a normal process, PMS is a problem, and that a specialist should be consulted when necessary. In addition, women should be supported and educated about healthy living and the necessary interventions to alleviate premenstrual symptoms before using analgesics, which is the first method used to cope with premenstrual symptoms. Nurses can also benefit from non-pharmacological methods to reduce the effects of premenstrual symptoms, support women in continuing their daily activities, increase their quality of life, and also provide pain and stress management. They can recommend non-pharmacological methods such as reflexology, meditation, yoga, distraction, imagination, massage, showering, hot and cold application, and relaxation techniques such as adequate sleep and rest.

ELIGIBILITY:
Inclusion Criteria Women who are 18 years of age or older, No communication problems, Scoring 111 and above on the Premenstrual Syndrome Scale, Having regular menstruation for the last six months, Having a menstrual cycle of 22-35 days, Having a menstrual period of no longer than 7 days, Not receiving medical or surgical treatment for PMS, Having no other gynecological problems, Having no psychiatric problems, Women who have no chronic illness in the last three months and have not undergone any gynecological surgery

Exclusion Criteria Women who score 110 or less on the Premenstrual Syndrome Scale, Women who are pregnant, Women who use hormonal contraception (such as oral contraceptives and injections), Women who have another gynecological problem, Women who have psychiatric problems, Women who have ulcers, varicose veins, thrombus, phlebitis, ecchymosis, hematoma, infection on both feet, women with impaired skin integrity, and women who have a history of foot surgery will not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participation of women diagnosed with premenstrual syndrome is mandatory
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Symptoms | 7 months
  Evaluation with Premenstrual Syndrome Scale

SECONDARY OUTCOMES:
Pain situation | 7 months
  Evaluation with Visual Comparison Scale

OTHER OUTCOMES:
Quality of Life Status | 7 months
  Evaluation with Quality of Life Scale

CONTACTS AND LOCATIONS:
Overall Officials: melike dişsiz, PhD, Study Director — Saglik Bilimleri Universitesi

IPD SHARING:
Plan to Share IPD: No